CLINICAL TRIAL: NCT02879864
Title: Effect on Fatigue of Light (Lux) Therapy in Patients With Cancer
Acronym: EFFLUX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EFFLUX
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: fatigue; tiredness; luxo therapy; therapy by light
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light therapy (Experimental): Light therapy takes place in the patient's home the day following receipt of the equipment and for at least 7 days before the start of chemotherapy and according to current recommendations: daily exposure to a high intensity light (10,000 lux) in the morning at a time to be adapted to the patient according to his chronotype), for 30 minutes. Light therapy begins immediately after receipt of the luminometer. The total duration of daily outpatient therapy program is 6 months. A set of questionnaires evaluation of fatigue and quality of life will be given to the patient at the inclusion visit and at weeks 12 and 24. They will complete the same day or the day before, and / or before any chemotherapy. A follow-up visit will be performed 1 month after the end of therapy (week 28).
  Interventions: Device: light therapy
- usual care (Active Comparator): usual care in oncology: The patient will be taken care of according to local chemotherapy in routine care and the recommendations. A set of questionnaires evaluation of fatigue and quality of life will be given to the patient at baseline and at weeks 12 and 24. They will complete the same day or the day before, and / or chemotherapy before . A follow-up visit will be performed 1 month after the last visit (week 28). A set of questionnaires evaluation of fatigue and quality of life will be given to the patient and will complete the same day or the day before
  Interventions: Device: Usual care

INTERVENTIONS:
Device: light therapy — The light therapy, 6 month's program, is occurring at patient's home the day after device's reception and during at least 7 days before chemotherapy's beginning. The ambulatory light program is daily exposure to a high-intensity light (10,000 lux) in the morning, at a time adapted to the patient according to his chronotype for 30 minutes. The light source should be placed at eye level (distance of about 40 cm). A set of questionnaires evaluation of fatigue and quality of life will be given to the patient at baseline and at weeks 12 and 24, which will be completed the same day or the day before, and / or before any chemotherapy. These questionnaires will be also completed during the follow-up visit 1 month after the last visit (week 28).
  Arms: Light therapy
Device: Usual care — The patient will be taken care of according to local chemotherapy in routine care and the recommendations. A set of questionnaires evaluation of fatigue and quality of life will be given to the patient at baseline and at weeks 12 and 24. They will complete the same day or the day before, and / or chemotherapy before. A follow-up visit will be performed 1 month after the last visit (week 28). A set of questionnaires evaluation of fatigue and quality of life will be given to the patient and will complete the same day or the day before.
  Arms: usual care

SUMMARY:
Fatigue is a symptom most commonly associated with the diagnosis of cancer. Fatigue often appears before the diagnosis of cancer, is increasing during treatment with chemotherapy and persists for years after treatment in more than 35% of patients. Fatigue is the earliest and most important symptom described by cancer patients. Its prevalence in cancer chemotherapy patients is between 70 and 100%. Fatigue is more common to cancer patients and to the general population or other types of patients. Typically described as a lack of energy associated with mental disorders, fatigue related to cancer can be extremely debilitating. The causes are many, mainly including the cancer itself, side effects due to treatment, sleeplessness due to pain, anxiety or depression. The cancer-related fatigue has a negative and significant direct impact on all aspects of the patient's quality of life, especially the physical, social and behavioral. Despite the availability of certain treatments and the advanced biomedical research, fatigue remains an inevitable consequence of cancer and its treatment.

The therapeutic use of natural light in medicine dates back to the late nineteenth century. Its remarkable effect on the stimulation of the immune system and fight against infections caused the development of the first therapy techniques (also called luxthérapie) awarded in 1903 by the Nobel Prize in medicine and physiology. Light plays a fundamental role in the regulation of circadian rhythms and homeostatic. The mechanism of action passes through a path "non-visual" involving melanopsin ganglion cells located in the retina. Activation of the pineal gland (epiphysis) by melanopsin cells allows transduce information "shadow and light" in melatonin synthesis from serotonin. Today, the effectiveness of the therapy is well established for treating fatigue-related disorders such as chronic fatigue, seasonal depression or seasonal or non-certain sleep disorders and in which the melatonin metabolism is disturbed. Light therapy, by its mechanism of action, allows reprogramming "of the biological clock and improved synchronization of circadian rhythms.

DETAILED DESCRIPTION:
Hypotheses

Some studies have shown an inverse relationship between cancer-related fatigue and the time of exposure to natural light for cancer patients. This association suggests the existence of a vicious circle of side effects of chemotherapy (physical fatigue and moral), itself causing a decrease in outdoor activity and therefore a reduction of the light exposure time natural. This results in a strengthening of the initial patient's state of fatigue. In an interesting way, vitamin D synthesized in large part due to light plays a cancer protective role], especially in the prevention and treatment of pancreatic cancer for example. Furthermore and paradoxical way, the disruption of circadian rhythms is correlated to the development and tumor progression in vitro, in vivo tumor growth and incidence of cancer in humans.

Notoriously, the direct effect of light therapy on cancer-related fatigue has been little discussed in the literature. Data obtained from a small sample of patients indicate that light therapy improves quality of life by reducing fatigue in patients with breast cancer during chemotherapy. To date, There are no data on the effects of light therapy on cancer-related fatigue in general, patients treated with chemotherapy.

The purpose of this pilot study is to evaluate the role of light therapy on cancer-related fatigue in patients during the 6 months following initiation of first-line chemotherapy.

Primary objective

To assess the effects of daily therapy on fatigue of patients with locally advanced or metastatic cancer treated with chemotherapy.

secondary objective

Evaluate the impact of daily light therapy on quality of life, pain, anxiety and depression, tolerance of chemotherapy and medico-economic benefits.

ELIGIBILITY:
Inclusion Criteria:

* Cancer histologically or cytologically confirmed (regardless of type)
* Patient eligible for first-line chemotherapy
* Life expectancy> 3 months
* WHO PS ≤ 2
* Age ≥ 18 years
* Informed consent signed and dated
* Affiliation to a social security scheme

Exclusion Criteria:

* Macular degeneration
* Diabetic retinopathy
* Glaucoma
* untreated cataract
* Patient treated with vitamin D
* Psychiatric disorders (bipolar disorder, paranoia, schizophrenia)
* For patients with other comorbidities may indicate against-the practice of therapy: application specialist opinion (ophthalmologist or psychiatrist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of Tiredness: PIPER Score | Day 1, week 12, week 24 and week 28
  Tiredness: PIPER Score (main variable) (22 items targeted in 4 dimensions: behavioral tiredness / intensity, emotional, sensory and cognitive / mood)

SECONDARY OUTCOMES:
Assessment of change of Quality of life (EORTC-QLQ-C30 SCORE) | Day 1, week 12, week 24 and week 28
  Quality of life related to health: EORTC-QLQ-C30 (30 items targeted in 4 dimensions: the overall quality of life, fatigue, physical functioning and pain).
Assessment of change of Health General condition WHO SCORE | Day 1, week 12, week 24 and week 28
  General condition: WHO
Assessment of change of Pain SCORE | Day 1, week 12, week 24 and week 28
  Pain: BPI-Short Form (BPI-SF) and analgesic consumption
Assessment of change of Depression Scale | Day 1, week 12, week 24 and week 28
  Depression / Anxiety: scale of depression and anxiety (HADS)
Assessment of change of slumber | Day 1, week 12, week 24 and week 28
  Sleep: Pittsburgh questionnaire (PSQI)

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided